CLINICAL TRIAL: NCT02607631
Title: A Phase II Study of Pembrolizumab for Patients With Thymic Epithelial Tumor Who Progressed After at Least One Previous Regimen of Cisplatin-Containing Chemotherapy
Brief Title: A Study of Pembrolizumab for Patients With Thymic Epithelial Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-04-132-005
Record Dates: First submitted 2015-10-07; First posted 2015-11-18 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Thymic Epithelial Tumors
Keywords: Thymic epithelial tumors; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Pembrolizumab 200mg IV every 3 weeks until tumor progression or unacceptable toxicity
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — treated with Pembrolizumab 200 mg every 3 weeks

SUMMARY:
This is a Phase II single center, open-label, single arm study in patients with advanced thymic epithelial tumors after failure of cisplatin-based combination chemotherapy. Patients will be treated with Pembrolizumab 200 mg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Histologically proven thymic epithelial tumor (TET) patients
4. Inoperable or metastatic disease
5. More than one previous chemotherapy including at least one platinum-based regimen
6. At least one measurable lesion based on RECIST 1.1
7. Patients who could submit at least one unstained slide to evaluate the PD-L1 expression status (PD-L1 status, which is positive (expression > 1percent of tumor cells) or negative, is the prerequiste for the enrollment. If the submitted slides are unacceptable for the analysis for PD-L1 and there is no remained slide, the patient cannot be enrolled)
8. Have a performance status of 0 or 2 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in Table 1. Laboratory test must be performed within 10 days before date of treatment.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
4. Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
5. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
6. Has an active infection requiring systemic therapy.
7. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
8. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
9. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
10. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
11. Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
12. Has known active tuberculosis which was not treated
13. Has a known history of hypersensitivity to pemborolizumab
14. Has a treatment history wih mAb within 4 weeks prior to the first dose of trial treatment
15. Has had radiotherapy or chemotherapy within 14 days of the first does of trial treatment. Subjects who received radiotherapy >14 days prior to randomization must have completely recovered from any therapy related AEs/toxicities except peripheral neuropathy less than grade II
16. Has a known history of psychosis or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Response rate by RECIST 1.1 | 24 months
  complete response plus partial response as determined by RECIST 1.1

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  include safety profiles
Progression free survival | 24 months
  time from the on-study date to date of disease progression
Overall survival | 24 months
  time from the on-study date to death as a result of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Prof., Principal Investigator — Samsung Medical Center

REFERENCES:
- [Derived] Kim KH, Cho J, Ku BM, Koh J, Sun JM, Lee SH, Ahn JS, Cheon J, Min YJ, Park SH, Park K, Ahn MJ, Shin EC. The First-week Proliferative Response of Peripheral Blood PD-1+CD8+ T Cells Predicts the Response to Anti-PD-1 Therapy in Solid Tumors. Clin Cancer Res. 2019 Apr 1;25(7):2144-2154. doi: 10.1158/1078-0432.CCR-18-1449. Epub 2019 Jan 15. PMID 30647082